CLINICAL TRIAL: NCT03811340
Title: Female Patient Preferences Regarding Physician Gender; is There a Difference? A National Survey
Brief Title: Female Patient Preferences Regarding Physician Gender
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 18-113
Record Dates: First submitted 2019-01-10; First posted 2019-01-22 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-10

CONDITIONS: Female Patient Preference

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross sectional survey study to describe female patient preferences when choosing their OB/GYN and other providers.

DETAILED DESCRIPTION:
The American College of Obstetricians and Gynecologists (ACOG) published that as of 2009, 79.7% of the Obstetrics and Gynecology residents were female. Given the striking decline in male providers selecting OB/GYN in more recent years, it is critical to characterize patient preferences in the current environment.

Nevertheless, it is not clear that females have strong preferences regarding gender. We hope to better understand the influence of bias on physician gender in present day.

The purpose of this study is to describe female population preference based on physician gender and specialty.

The study will be conducted on an online platform distributed across the United States by the aid of SurveyMonkey® .

ELIGIBILITY:
Exclusion Criteria:

* Unwillingness to participate in the study
* Lack of access to the internet
* Non-English speaking

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female population residing in the USA
Sampling Method: Non-Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1000 responses from females across the U.S were expected
Groups:
- Survey Population: All women between 18 and 80 years of age residing in the USA
Period: Overall Study
Arm/Group | Survey Population
Started | 1105
Completed | 1015
Not Completed | 90
Not completed — subjects did not complete the survey. | 90

BASELINE CHARACTERISTICS:
Arm/Group | Survey Population
Number analyzed (Participants) | 1015
Age, Customized [Count of Participants; unit: Participants]
  18-30 | 339
  31-45 | 189
  46-60 | 373
  61-75 | 107
  >75 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1015
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic | 865
  Hispanic | 135
  Prefer not to answer | 13
  No response | 2
Region of Enrollment [Number; unit: participants]
  United States | 1015

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Female Respondents Having Their Preferences Based on Physician Gender for the OB/GYN Care
Description: Proportion of female respondents whose responses are "Male physician" or "Female physician" over "No preference" for the question 15, "For my obstetrician/gynecologist, overall I would prefer a..."
Time Frame: During a 10 minute period of completing the survey electronically
Measure: Count of Participants; unit: Participants
Arm/Group | Survey Population
Number analyzed (Participants) | 1015
Participants
  Female physician | 667
  Male physician | 87
  No preference | 261

2. Primary Outcome: Proportion of Female Respondents Having Their Preferences Based on Physician Gender for the Primary Care Physician
Description: Proportion of female respondents whose responses are "Male physician" or "Female physician" over "No preference" for the question 16, "For my primary care physician, overall I would prefer a..."
Time Frame: During a 10 minute period of completing the survey electronically
Measure: Count of Participants; unit: Participants
Arm/Group | Survey Population
Number analyzed (Participants) | 1015
Participants
  Female physician preferred | 473
  Male physician preferred | 102
  No preference | 440

ADVERSE EVENTS:
Time Frame: During a 10 minute period of completing the survey electronically
Arm/Group | Survey Population
All-Cause Mortality (participants affected / at risk) | 0/1015
Serious Adverse Events (participants affected / at risk) | 0/1015
Other Adverse Events (participants affected / at risk) | 0/1015

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT03811340/Prot_SAP_000.pdf